CLINICAL TRIAL: NCT03076398
Title: Feasibility Study and Prototype Computerised Program Development of Anaesthesia Electronic Medical Record
Brief Title: Development of Anaesthesia Electronic Medical Record
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Phongthara Vichitvejpaisal, Professor, Siriraj Hospital
Other Study IDs: Si 140/2016
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Normally, anaesthesia personnel make a record patients' information during the surgical procedure. Pre and post-operatively, they visit patients to make sure that their customers are well informed regarding the whole process and satisfied with the service as well as any complications that might be existed.

The investigators would like to develop an anaesthesia electronic medical record at the point of care. The objectives are to record peri-operative patients' information in a real-time fashion, manage all administrative tasks as annual reports, and operate data as search engine for research and educational purpose.

DETAILED DESCRIPTION:
Department of Anaesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University provides services to patients undergoing operative procedures in many fields; such as Traumatic surgery, Orthopaedics surgery, Eye surgery, Ear, Nose and Throat surgery, Plastics surgery, Cardio-thoracic surgery, Neurosurgery, General surgery, Urological surgery, Head and Neck surgery, Paediatric surgery, Obstetrics surgery, Gynaecological surgery, Electro-convulsive therapy, Radiological services, Endoscopic centre, Intensive Care Unit, Acute Pain service, Pain Clinic and Pre Anaesthesia Assessment Centre.

Normally, anaesthesia personnel make a patient information record during the surgical procedure. Pre and post-operatively, they visit patients to make sure that their customers are well informed regarding the whole process and satisfied with the service as well as any complications that might be existed.

The patient data, a crucial document for both medical and official terms, has been developed and improved continuously by the department. Daily, about 250 informations are transferred from paper-pencil to electronic, computerised format for statistical purpose and further reference. Still, the department has to face the data problem in many aspects.

1. Daily, an abundant of information needs to be transferred to computer by non-medical personnel. This results in time consuming, data loss and piles of document.
2. Unclear peri-operative handwriting of medical or technical terms, particularly on copied files results in untrustworthy and disgraceful of patients' evidence.
3. Scanned files results in difficulties of data retrieval for assignments in research, education, administrative policy and finance. Consequently, a hospital becomes an unfaithful and treacherous organisation.

The investigators would like to develop an anaesthesia electronic medical record at the point of care. The objectives are to record peri-operative patients' information in a real-time fashion, manage all administrative tasks as annual reports, and operate data as search engine for research and educational purpose.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing anaesthesia

Exclusion Criteria:

* N/A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing general or regional anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 397 (Estimated)
Dates: Start 2015-02-19 (Actual); Primary Completion 2017-04-19 (Estimated); Study Completion 2017-04-19 (Estimated)

PRIMARY OUTCOMES:
Anaesthesia Electronic Medical Record | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Shayakul, Study Chair — Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand
Locations (1):
- Phongthara Vichitvejpaisal, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No